CLINICAL TRIAL: NCT02971241
Title: Intergenerational Mobile Technology Opportunities Program (IMTOP) in Taiwan
Brief Title: Intergenerational mHealth Diabetes Program OPPORTUNITIES PROGRAM IN TAIWAN
Acronym: IMTOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Taipei Fubon Bank Charity Foundation (Unknown); Taichung Tzu Chi Hospital (Other); Hualien Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Shinyi Wu, Associate Professor, University of Southern California
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UP-15-00270
Record Dates: First submitted 2016-11-19; First posted 2016-11-22 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Integeneration; Mobile technology; Chronic disease management; Diabetes self-management
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Quasi-experimental wait-listed control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate intervention group (Experimental): A randomized, waitlist controlled trial with three hundred fifty older adult subjects with type 2 diabetes and 280 young adult subjects will be conducted in Taipei Tzu Chi Hospital and Hualien Tzu Chi Hospital in Taiwan. The patients who are randomized to the immediate intervention group will be assigned to the training course as soon as a course is available.
  The intervention is a 12-week program which consists of 8-week training sessions followed by 4-week consultation service for technical support. Both will be provided by the young volunteers with a lead instructor.
  Interventions: Behavioral: Intergenerational Mobile Technology Opportunities Program
- Waitlist control group (Other): The patients randomized to the waitlist control group will need to wait for four months to serve as no intervention control, and then assigned to the training course.
  Interventions: Behavioral: Intergenerational Mobile Technology Opportunities Program

INTERVENTIONS:
Behavioral: Intergenerational Mobile Technology Opportunities Program — The themes of the 8-week training session are designed based on the objectives of IMTOP: 1) teach skills of tablet use and diabetes self-management behavior tracking app, 2) introduce online community communication to decrease social isolation and obtain social support from family and friends, young volunteers, health care providers, and diabetes peers who have similar condition/interest/ or disease), 3) teach diabetes self-management knowledge and skills based on the evidence-based Chronic Disease Self-Management Program; and 4) teach mobile technology application to healthcare access and daily needs (i.e., online appointment, online refill, appointment reminder, online health information, online training videos, and virtual classes such as e-newspaper, e-books, related sites, apps).

SUMMARY:
The primary purpose of the study is to understand the potential of mobile computing technology to improve chronic disease self-management, quality of life, and health outcomes of older adults to prevent or alleviate future disabilities. Thus, the study will design, develop, and test an intervention to motivate and train seniors to use the technology, and conduct a trial to evaluate its effect. This innovative intervention will deploy young generation (age 18 to 30) volunteers to provide mobile technology training, access, and support to older adults (aged 55 and above) with type 2 diabetes in Taiwan. Hence, a secondary purpose of the study is to understand the effects of the volunteering experience on the values, characters, and health awareness in the young generation. This program, called the Intergenerational Mobile Technology Opportunities Program (IMTOP), will help older adults with type 2 diabetes acquire skills to use the Internet, World Wide Web (WWW), applications (or "apps"), and basic computing via mobile tablet devices. These skills will give participants access to resources and tools to improve health and mental health, reduce social isolation, and increase social engagement, as well as meet their individual life goals. The course will use young volunteers to deliver the tablet training. The training course will be offered as small-group sessions over an 8-week period (for up to 16 hours of training) at a hospital site, plus young volunteers' technical support and problem solving for up to 4 weeks after the training sessions are completed. Using college students to serve as volunteer trainers for teaching mobile technology, the research also aims to understand not only how the intergenerational interactions help the older adults learn the technology and improve health, but also how the tutoring experiences make impact on the young adults' skills and perspectives that will help them in their future careers and in the development of their characters. This research study will recruit three hundred fifty (350) patients from the collaborating hospitals, including two hundred fifty (250) patients from Taipei Tzu Chi Hospital and one hundred (100) patients from Hualien Tzu Chi Hospital. An estimate of 140 students in colleges and universities in Taiwan (100 volunteers in Taipei hospital and 40 volunteers in Hualien hospital) between the age of 18 and 30 will be recruited to serve as volunteer instructors to teach older adults to use tablets and to provide technical support services. Moreover, another group of 140 young adults, also age 18 to 30, will be recruited from universities to serve as the comparison group to the volunteers in intervention group. The course objectives are to guide older patients with Type 2 diabetes to use technology to obtain diabetes-related medical information, learn to record and control their physiological data via technology, promote intergenerational communication, enhance the convenience in life, and improve social life and mental health through technology tools such as the Internet, social media, online health education resources, instructional videos and so on. It is hoped to further slow down degradation, promote health and prolong life.

DETAILED DESCRIPTION:
The research design is a randomized waitlist control trial. Patients will be randomly assigned to the immediate intervention group or 4-month waitlist control group. The former will immediately join the tablet computer courses, while the later will wait for four (4) months before starting their courses. The follow-up period for patients will be one (1) year after the start of courses. Patient assessments will include baseline and follow-up assessments of health behaviors, functional status, health conditions, and social interactions and engagements, plus technology use and acceptance. Baseline assessment will be conducted at recruitment for all patients, and for waitlist control group again at the beginning of the course. Follow-up assessments will be conducted at four (4) months, eight (8) months, and twelve (12) months after the start date of the courses. Young volunteers will also be assessed to understand their experiences in the volunteering services and any impact from this experience. The assessments will be conducted at the baseline, during the courses, and two (2) months and four (4) months after the beginning of the courses. In addition, a group of 140 young adults will be recruited from universities to serve as the comparison group and will be asked to complete the assessment survey at baseline, two (2) months, and four (4) months later.

For older adults:

Patients who meet inclusion criteria will be referred by doctors in the metabolism and endocrinology department of the two hospitals to recruiters and will be randomly assigned to immediate intervention group and waitlist control group. The aim of the comparison is to assess the potential effects of mobile technology program with intergenerational interaction on patients' technology use, self-efficacy, self-management behavior, and social engagement, and whether it results in less social isolation and health care utilization, improved health and mental health status, and greater quality of life.

Recruitment procedure:

1. Tzu Chi diabetes health educators will recruit patients with type 2 diabetes and screen them for eligibility. The health educators will complete a patient contact card for each patient that they screen for eligibility. If eligible, the health educators will explain the study to the patients and ask for their interest to participate. Interested patients will be referred to an IMTOP study recruiter. The recruiter will collect all patient contact cards and completed screeners from the health educators.
2. The study recruiters on site in the hospital will obtain the informed consent from the eligible and interested patients. When the patients sign the study consent, the recruiter will write on the patient contact card the patient ID next to Study Participation Status - Enrolled, and complete the patient contact card.
3. The recruiter will then conduct the baseline interview. Baseline interview can be done face to face or via telephone if patient prefers.
4. Patient's study group (immediate intervention or wait list control group) will be randomly assigned at the study's Qualtrics database after baseline interview is complete.
5. All recruitment paper, if any, will be sent to the project manager to file on a locked cabinet.
6. The patients who are randomized to the immediate intervention group will be assigned to the training course as soon as a course is available. The patients randomized to the waitlist control group will need to wait for six months to serve as no intervention control, and then assigned to the training course.

Description of intervention:

The intervention is a 12-week program which consists of 8-week training sessions followed by 4-week consultation service for technical support. Both will be provided by the young volunteers. The themes of the 8-week training session are designed based on the objectives of IMTOP: 1) teach skills of tablet use, 2) introduce online community communication to decrease social isolation and obtain social support from family and friends, young volunteers, health care providers, and diabetes peers who have similar condition/interest/ or disease), 3) teach diabetes self-management knowledge and skills based on the evidence-based Chronic Disease Self-Management Program; and 4) teach mobile technology application to healthcare access and daily needs (i.e., online appointment, online refill, appointment reminder, online health information, online training videos, and virtual classes such as e-newspaper, e-books, related sites, apps).

Moreover, the enrolled older adults will be invited to use a diabetes self-management behavior tracking app developed by the research team. The app is designed to encourage diabetes patients to regularly record their diet, physical activity, water consumption, medication adherence, blood sugar readings, and blood pressure readings. The data will be used for our research analysis to understand to what extent the older adults use the app and whether regular recording has impact on the outcome measures.

The 4-week consultation service post the 8-week training course is intended as additional support for the older adults who encounter technical issues when using the tablet on their own. To receive the technical support, the older adults shall call the study hotline or post their questions on the study website to explain the technical issues. The research staff will find a study volunteer to address the technical issues.

During the training sessions in the classroom, the research team may audiotape, videotape, or take photos to record classroom interactions between older adults and young volunteers. The recordings will be no more than half of the 8 sessions and each time we may videotape up to 90-min per session. The purposes are for quality improvement of the IMTOP program, for research analyses at the aggregate level, and for dissemination of the program. The participants have the rights to decide whether to be taped or photographed. They may indicate their decision on the consent form or by telling the recorder/photographer at the time of the taping/photo shooting.

Accrual and baseline data collection:

University of Southern California (USC) research team will prepare enrollment packages (including an information sheet, the screener, the patient contact card, the consent form, HIPPA form and a 40-minute baseline survey). Health educators employed by two Tzu Chi Hospitals will help enroll and consent eligible patients. Participating patients will be asked to sign the HIPPA authorization form to release their medical records in hospitals. Consenting patients will be invited to take baseline survey through an interview with a study interviewer, either in-person or by phone based on patient's preference. When baseline survey is completed, patients will be randomly assigned to intervention group and wait-list control group.

Follow-up survey: For immediate intervention patients, 4-month, 8-month, and 12-month follow-up surveys will be administered via telephone by part-time interviewers employed for the study by the hospitals. For wait-list control group patients, 4-month, 8-month, 12-month, and 16-month follow-up surveys will be administered via telephone by the part-time interviewers. Study data will be obtained from patients' self-report on study assessments, study tracking records such as the training course attendance, and patients' medical records pertaining to diabetes care and healthcare utilizations in Taipei and Hualien Tzu Chi Hospitals. Self-report data collected from patients include demographic characteristics, physical health and mental health status, self-management behaviors, health care utilization, health literacy, self-efficacy, social engagement, and quality of life. The study assessments and study tracking records will be conducted exclusively for research purposes.

For young volunteers:

Accrual and baseline data collection:

IMTOP research staff and employees (such as diabetes health educators) of the Taipei and Hualien Tzu Chi Hospitals will distribute young volunteer recruitment flyers to officer of student affairs and faculty at various universities nearby the study sties. The IMTOP research staff will also arrange meetings at university campuses to introduce the study and call for volunteers. The study information and the call for volunteers will be disseminated campus wide two months prior to each IMTOP training term starts.

Young adults who are interested in participating in the study as volunteer instructors for the training course will sign up at the study website IMTOP.usc.edu. The sign-up section of the website will explicitly show the language that enrollment in the study means a volunteer is not only serving as an instructor but also as a research participant. To complete the sign up will require acknowledgment of the dual roles. There will be a study hotline number shown on the recruitment flyer for interested young adults to get more information about the study and for sign-up. The research staff will contact those young adults who meet the study inclusion criteria for an interview to clarify the job responsibilities and the expectations. Those who agree to meet the expectations will be invited to attend the two-day training workshop (described below).

On the day of the training workshop, the young adults will be asked to consent for their study participation and to complete the study baseline. Then they will be accepted for the study enrollment as young volunteers. The target recruitment is 140 volunteers.

USC research team will prepare the enrollment package (including the recruitment flyer, the sign-up form, the consent form, and a 40-minute self-administered baseline survey). The sign-up and the consent form will be available via the study website IMTOP.usc.edu. The self-administered surveys will be available on qualtrics website via a web link in the study website.

Orientation workshop:

USC research team will provide two orientation workshops for enrolled volunteers to learn skills and knowledge for delivering the intervention service. The topics of orientation workshops include young volunteers' role and responsibilities in the IMTOP research project, knowledge of aging process, motivational interviewing skills, problem solving skills, empathy, communication with older adults, and introduction of the 8-week training curriculum and the 4-week technical support.

Volunteering services:

After the orientation workshop is successfully completed, young volunteers will be assigned to be one of about 4 instructing volunteers to provide the tablet training for a group of approximately 10 older adults with type 2 diabetes. The training course is 2 hours per session and 1 session per week for 8 weeks long. In each session, there is a prepared course material for the volunteers to deliver to the older adults, such as use of web browsers, application of social media, and online supporting materials for the older adults to learn mobile technology for their self-management to improve health and quality of life. After the 8-week training period, the young volunteers will provide 4-week technical support for the diabetes outpatients via phone or mobile device.

During the tablet training sessions in the classroom, the research team may audiotape, videotape, or take photos to record classroom interactions between older adults and young volunteers. The recordings will be no more than half of the 8 sessions and each time we may videotape up to 120-min per session. The purposes are for quality improvement of the IMTOP program, for research analyses at the aggregate level, and for dissemination of the program. The participants have the rights to decide whether to be taped or photographed. They may indicate their decision on the consent form or by telling the recorder/photographer at the time of the taping/photo shooting.

Baseline and follow-up survey:

The enrolled young volunteers will be asked to complete the self-administered online surveys at baseline and at 2-month and 4-month follow up. That is, the baseline will be completed prior to the intervention. The 2-month follow-up will be completed immediately after the 8-week training course. The 4-month follow-up will be completed one month after the 4-week technical support period. The survey will collect data about demographic characteristics, level of empathy, citizenship behavior, time management skills, altruism value, purpose of life, and career development. In addition, the young volunteers will be asked to take turn in recording the class log, including the class attendance, materials taught, Q&A, any difficulty or questions in delivering the curriculum, and other relevant observations or issues. Additionally, once a month for a total of three times, once in week 4 and once in week 8 during the 8-week course, plus once in the end of the 4-week technical support, they will be asked to write a short reflection of their volunteering experience. These study assessments and study tracking records will be conducted exclusively for research purposes.

For young adult comparison group:

A group of 140 young adults similar to the young volunteers will be recruited from universities through information meetings held by the research staff in collaboration with officer of student affairs and faculty at various universities. They will not be randomized, but instead they will be deliberately recruited to be the comparison group that matches with the young volunteer group on the bases of age range, college attendance and major, and location of the schools. These young adults will be informed to serve as the comparison group for the study. Once consented, they will be directed to answer the same self-administered online surveys at baseline and at 2-month and 4-month follow up.

Data Storage and Confidentiality:

1. All questionnaires completed electronically via the web-based survey company qualtrics, license available through the USC Information Technology Services (http://www.usc.edu/its/qualtrics/), will be kept in the secure website of qualtrics and then downloaded into a centralized database located in the USC School of Social Work. The following links show privacy, acceptable use, and security statements provided by qualtrics:

   http://www.qualtrics.com/privacy-statement/ http://www.qualtrics.com/acceptable-use-statement/ http://www.qualtrics.com/security-statement/
2. Data collected on the study website IMTOP.usc.edu will be stored in secure and password protected website at Amazon Cloud Drive, and then downloaded into a centralized database located in the USC School of Social Work.
3. A password protected secure computer file linking identifying information and the subject study ID will be securely maintained under control of Dr. Wu and the study Data Analyst in the School of Social Work.
4. All study data files will only contain subject IDs, not identifying information.
5. Analysis and publication of the data will employ procedures making it impossible to identify individuals.
6. After completion of the study, identifiable data such as video tapes will be destroyed, but the remaining data will be retained at the researchers discretion and may be used in future research studies. ..
7. All study investigators and staff have already or will complete the USC IRB and required HIPAA certification course.

Hardcopy study data will be kept in the secure location in the USC School of Social Work or in a designated locked cabinet in the collaborating Tzu Chi hospitals for a period of 5 years following study completion, after which it will be destroyed. Study tracking data will also be kept on a secure, password protected, web-site maintained by the School of Social Work within the Hamovitch Research Center.

RISK/BENEFIT ASSESSMENT

Potential Risks:

There are no anticipated risks to subjects' participation in this study. The tablet training program takes place in Taipei or Hualien Tzu Chi Hospital. Subjects' participation in the program may involve normal risks in transportation to attend the training sessions. Frequency and intensity of training sessions might cause them certain level of anxiety and discomfort, such as soreness in eye.

As the study subjects will also participate in the study surveys, some of the survey questions may make them uncomfortable or concerned, but they can choose not to answer any questions they do not wish to answer. Participating in research may involve a loss of privacy, but all of the information the subjects provide will be kept confidential. The possibility of a breach of privacy to occur is very low but will exist as long as we hold the data.

All participants will be advised that they are free not to use the technology and not to answer any questions that make them uncomfortable. However, in previous studies of depressed patients, distress resulting from interviews and questionnaires has been minimal. Subjects may experience inconvenience and time costs associated with using technology and completing study interviews; however, all interventions and interviews are completely voluntary and will be conducted at the participant' convenience.

The technology intervention does not expose patients to additional or unusual medications or side effects.

Although all efforts will be made to protect patient confidentiality, those patients who experience critical clinical events (e.g., hypoglycemia) during the study training sessions or those who are likely victims of abuse may experience loss of confidentiality as study staff will be required to report these events to the subject's physician for appropriate safety measures to be taken.

Risk Classification:

The risks of this study are consistent with the HHS/FDA Regulations definition of minimal risk.

Protection Against Risks:

The study PIs and the project manger who has a gerontology and public health background will train the study recruiters, interviewers, and young volunteers to handle distressed or potentially at risk patients during recruitment, intervention, and assessment. The recruiters, interviewers, and young volunteers will request permission from distressed subjects to notify their physician so that they may be assessed and treated as necessary. In the case of emergengy, the recruiters, interviewers, and young volunteers will inform the patient of the immediate need to notify the patient's physician, even without his or her permission, so that these providers may take appropriate action to ensure patient safety. This will involve using usual clinic channels to have the patient urgently evaluated and and appropriate disposition arranged (including possible transport to Emergency Department in Taipei and Hualien Tzu Chi Hospitals). The study principal investigator in the local site will be available by cellular phone and will also be notified of emergency patients in order to to ensure timely assessment and treatment by a physician.

Data Safety Monitoring Plan:

All assessment data will be entered into a centralized database located in the USC School of Social Work. Study patients will be identified by a unique study code number, the identity of which will be known only to the study personnel with direct responsibility for providing patient data. The database will be password protected against non-project personnel and backed up weekly. This removes patient-identifiable data from the files. The data manager and biostatistician will create a series of databases in Excel and SAS, so that they can analyze the initial data as it comes in to ensure proper patient recruitment, track progress of the study, and perform data checks and cleaning. All baseline and follow-up data, including responses to the screener questionnaire, will be entered on qualtrics web-based survey system through tablets or other computer devices onsite. The data will be identified by the patient's study ID code. This data will be transmitted either wirelessly, through third or forth generation mobile telecommunications, or through the local network connection in real time to the qualtrics server as data is entered by recruiters on the computer devices, which has been loaded with the requisite software and encryption system. The transmitted data will be encrypted using HIPAA-compliant encryption and password protected. If there is poor wireless connection or mobile telecommunication transmission is not possible, recruiters will enter baseline and follow-up data on paper forms. All forms will be checked for completeness by the qualtric systems or, if paper, by the study coordinator before being sent to the project manager. The project manager will review and double-check all of the forms to be sure they are completed and readable. For data on paper forms, data will be entered singly using SAS (SAS Institute Inc., SAS Campus Drive, Cary, NC) full screen editor (FSEDIT) into SAS database system with back-up copy and hard copy kept in secure locked file cabinet in the SSW. For data on the qualtrics server, data would be downloaded onto local sites into the SAS database system with back-up copy password-protected. Accuracy of data entry will be ensured by an internal program with FSEDIT for range and logic check, and by a comparison between printouts and the handwritten data forms. To assist in monitoring the study, periodic reports will be generated using graphs and tables summarizing the status of subject recruitment and data collection. Missing data will be routinely rectified. SAS will also be used to analyze the data and generate all statistical reports. Data on the qualtrics server and the project website will be destroyed at the end of the study.

Potential Benefits to the Subject and/or Society:

Direct benefits to patients who participate IMTOP study include learning: 1) skills of tablet use, 2) online community communication with family and friends, young volunteers, health care providers, and diabetes peers who have similar condition/interest/ or disease, 3) diabetes self-management knowledge and skills; and 4) mobile technology application to health access and daily needs (i.e., online appointment, online refill, appointment reminder, online health information, online training videos, and virtual classes such as e-newspaper, e-books, related sites, apps) at no or minimal out-of-pocket cost (e.g., transportation cost to attend the training course). There is a potential of improving the flow of communication between these patients and their health educators as well as physicians through using mobile technology. Self-management knowledge and behaviors will improve among them. Those patients in the waitlist control group may also experience benefits due to the raised levels of awareness of self-management, and later experience the potential benefits associated with the tablet training intervention. The potential benefit to society is that IMTOP intervention is likely to create an approach to improve self-management behaviors, health outcomes, and quality of life in patients with type 2 diabetes. In addition, with improvement in self-monitoring behavior among older diabetes patients and raised levels of health awareness among young volunteers, medical expenses of diabetes care by the government might decrease, which benefits the society as a whole.

Alternatives to Participation:

Refusal to participate will not negatively impact older adults' diabetes care or their access to usually available health services. If patients are interested in learning more about diabetes self-management skills, but do not wish to participate in the study, written educational materials in Chinese will be available.

Refusal to participate among young adults, either in the volunteering group or in the comparison group, also will not have any negative impact on the younger adults. They can request to receive a copy of written educational materials in Chinese for future diabetes prevention.

Risk/Benefit Relationship:

The potential benefits to participants are greater than the risks associated with participation. The physical, psychological, social, and legal risks to patients with type 2 diabetes are minimal. IMTOP study aims to improve their health outcomes and quality of life. In addition, the intergenerational interactions could be a motivator for them to learn the technology to enhance their skills of self-management, which may result in improved health and decreased cost of medical care as a whole.

For young volunteers, the risk is negligible but the focus of intergenerational interactions could potentially improve their communication with and empathy for older adults, increase awareness of self-care and disease prevention, build health-focused values of life style, and shape future career choice.

For young adults in the comparison group, although both risk and benefit are minimal, they may feel a sense of pride through their contribution to research.

ELIGIBILITY:
Inclusion Criteria:

Older adult subjects inclusion criteria are:

* current Taipei or Hualien Tzu Chi patients
* aged equal to or greater than 55 years
* having a current diagnosis of type 2 diabetes mellitus with duration of diagnosis at least 6 months
* having the ability of reading Chinese newspaper
* normal eye-hand coordination
* being able to regularly attend the IMTOP training course
* understanding Mandarin (listening, speaking, reading, and writing).
* having a working telephone at home or a cellular phone.

Younger adult subjects inclusion criteria are:

* age between 18 and 30
* having basic levels of verbal, interpersonal communication, and computer skills and commitment in voluntary works for approximately 50 hours during the period of intervention.

Exclusion Criteria:

Older adult subjects exclusion criteria are:

* a score of 2 or greater on the CAGE 4M alcohol assessment;
* having schizophrenia, schizoaffective disorder, manic-depressive, or needing lithium;
* cognitive impairment precluding ability to give informed consent or participating in the intervention, i.e., SPMSQ score of 4 or more errors.

Younger adult subjects exclusion criteria are:

* age less than 18 or above 30
* being unfamiliar with computer
* being unable to commit 50 hours during the period of intervention

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 617 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Patient survey | One year
  The survey collects data from patients include demographic characteristics, relationship with children and grandchildren, physical health (IADL) and mental health status, self-management behaviors, health care utilization and satisfaction, health literacy, self-efficacy, usage of app, social engagement, attitudes toward young adults and quality of life.
Young students survey | Four month
  The survey will collect data about demographic characteristics, level of empathy, citizenship behavior, time management skills, altruism value, purpose of life, attitudes toward older adults, relationship with grandparents and career development.

CONTACTS AND LOCATIONS:
Overall Officials: Shinyi Wu, PhD, Principal Investigator — University of Southern California
Locations (2):
- Taiwan (2):
  - HualienTzu Chi Hospital, Hualien City
  - Taipei Tzu Chi Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] International Diabetes Federation (2013). Diabetes: Facts and Figures. Retrieved from http://www.idf.org/worlddiabetesday/toolkit/gp/facts-figures Santos-Longhurst, A. (2014). Type 2 Diabetes Statistics and Facts. Retrieved from http://www.healthline.com/health/type-2-diabetes/statistics#2 Gregg, E. W., Mangione, C. M., Cauley, J. A., Thompson, T. J., Schwartz, A. V., Ensrud, K. E., & Nevitt, M. C. (2002). Diabetes and incidence of functional disability in older women. Diabetes Care, 25(1), 61-67. Gregg, E. W., Breckles, G. L. A., Williamson, D. E., Leveille, S. G., Langlois, J. A., Engelgau, M. M., Venkat Narayan, K. M. (2000). Diabetes and physical disability among older U.S. adults. Diabetes Care, 23(9), 1272-1277. Gregg, E. W., Breckles, G. L. A., Williamson, D. E., Leveille, S. G., Langlois, J. A., Engelgau, M. M., Venkat Narayan, K. M. (2000). Diabetes and physical disability among older U.S. adults. Diabetes Care, 23(9), 1272-1277. Glasgow, R. E., Kurz, D., King, D., Faber, A. J., Halterman, E., Woolley, T. Toobert, D. J., Strycker, L. A., Estabrooks, P. A., Osuna, D., & Ritzwoller, D. (2012). Twelve-month outcomes of an internet-based diabetes self-management support program. Patient Education and Counseling, 87, 81-92 Yo, N. C. (2014). One in every ten people is living with diabetes mellitus. Retrieved from http://www.tpuca.org/news_list/show/316.html World People News. (2014). Diabetes has been ranked as the fourth leading causes of death in Taiwan. Retrieved from http://www.worldpeoplenews.com/category/2/6 Ministry of Health and Welfare. (2014). Diabetes shared network. Retrieved from http://www.tpuca.org/news_list/show/316.html